CLINICAL TRIAL: NCT05320653
Title: Nutritional and Metabolic Characteristics of Critically Ill Patients Admitted for Severe Toxidermia
Brief Title: Nutritional and Metabolic Management of Toxidermia Patients Requiring Intensive Care (TEN Metabolism)
Acronym: TEN metabolism
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Mette M Berger, Prof.Hon., Centre Hospitalier Universitaire Vaudois
Other Study IDs: CER-2018-2268
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Stevens-Johnson Syndrome Toxic Epidermal Necrolysis Spectrum
Keywords: Critical care; Metabolism; Nutrition; Protein
MeSH Terms: conditions — Stevens-Johnson Syndrome | interventions — Nutrition Therapy; Parenteral Nutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 31 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Dietary Supplement: Medical nutrition — Nutrition therapy of the critically ill patients
  Other Names: enteral, oral and parenteral nutrition

SUMMARY:
Retrospective observational cohort study including all patients admitted for toxidermia (Lyell syndrome, Stevens-Johnson Syndrome (SJS), or other extensive skin destruction) to the Burn unit of the adult ICU of the Lausanne burn center between 2006 and 2020.

Inclusion criteria: age >18 years and admission to the burn-ICU for toxidermia whatever body surface affected.

Exclusion criteria: to have declined access to the medical record, a stay shorter than 24 hours, and major burns. The observation period will be limited to the first 31 days of the ICU stay.

All variables related to nutritional and metabolic management will be recorded

DETAILED DESCRIPTION:
There are yet no description of the metabolic characteristics of patients admitted for Toxic epidermal necrolysis (TEN) or Stevens-Johnson Syndrome (SJS) which are a rare condition, often assimilated to major burns in terms of metabolic requirements. We will conduct a retrospective observational cohort study including all patients admitted for toxidermia (general term including TEN or Lyell syndrome, SJS, and other extensive skin destruction) to the Burn unit of the adult ICU of the Lausanne burn center between 2006 and 2020. The primary outcome will be compliance with the ICU's feeding protocol (feeding route, early start of enteral feeding, ), and secondary outcomes will include the adequacy of energy and protein delivery, and use of indirect calorimetry, and the comparison with both general and burn critically ill patients from prior studies in the ICU.

Inclusion criteria: age >18 years and admission to the burn-ICU for toxidermia whatever body surface affected.

Exclusion criteria: to have declined access to the medical record, and a stay shorter than 24hours, and major burns. The observation period will be limited to the first 31 days of the ICU stay.

The recorded variables will include demographic characteristics, severity scores (SAPSII, SCORe of Toxic Epidermal Necrosis (SCORTEN for SJS/TEN), Nutrition risk screening (NRS) score), body surface area (BSA) affected by the disease, fluid intakes and balance (exudate volume estimation not included) of the first 10 days, body weight during the stay, renal function, length of mechanical ventilation and of ICU stay. Nutritional variables include the route of feeding, the 24hr energy prescription and delivery, protein, glucose, and lipid intakes, propofol, insulin, indirect calorimetry (IC) studies. Laboratory blood results include glucose, prealbumin, albumin, C-reactive protein (CRP), triglycerides, creatinine, and trace elements (Cu, Se, Zn).

Descriptive statistics: Wilcoxon rank test, while Chi2 test, changes over time with one-way ANOVA .

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* admission to the burn-ICU

Exclusion Criteria:

* declined access to the medical record
* stay shorter than 24hours

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Cohort of all patients admitted for SJS/TEN and other toxidermia
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Compliance with ICU feeding protocol | ICU stay, but maximum 30 days
  Proportion of ICU days with covered needs

SECONDARY OUTCOMES:
Protein delivery | ICU stay but maximum 30 days
  Delivery of at least 1.1 g/kg day of protein
Energy delivery | ICU stay but maximum 30 days
  Delivery of at least 25 kcal/kg/day

CONTACTS AND LOCATIONS:
Overall Officials: Eckert Philippe, MD, Study Director — Université de Lausanne, Director of the ICU

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karakus M, Pantet O, Charriere M, Favre D, Gaide O, Berger MM. Nutritional and metabolic characteristics of critically ill patients admitted for severe toxidermia. Clin Nutr. 2023 Jun;42(6):859-868. doi: 10.1016/j.clnu.2023.04.006. Epub 2023 Apr 8. PMID 37086614